CLINICAL TRIAL: NCT04510402
Title: Phase I/II Trial (Safety and Dosing) of Povidone-iodine (PVP-I) Nasal Swab For Preventing COVID-19 Spread in Healthy Subjects
Brief Title: Phase I/II Trial of Povidone-iodine (PVP-I) Nasal Swab For Preventing COVID-19 Spread in Healthy Subjects
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: 3M (Industry)
Responsible Party: Principal Investigator, Raymond Manohar Anchan, M.D.,Ph.D., Assistant Professor HMS, Associate Gynecologist, BWH, Brigham and Women's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2020p002323
Record Dates: First submitted 2020-08-10; First posted 2020-08-12 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Covid19; Povidone Iodine Adverse Reaction
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Fifty healthy volunteers to use single application or double application of PVP-I nasal swabs and assess for safety and tolerability
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Safety Analysis (Experimental): Evaluate safety of PVP-I nasal swabs single daily application
  Interventions: Drug: Povidine iodine nasal swabs
- Tolerability analysis (Experimental): Investigate the dosing of PVP-I nasal swabs daily single dosing versus double dosing
  Interventions: Drug: Povidine iodine nasal swabs

INTERVENTIONS:
Drug: Povidine iodine nasal swabs — Daily versus twice daily nasal application

SUMMARY:
Title: Phase I/II Trial (Safety and Dosing) of Povidone-iodine (PVP-I) Nasal Swab For Preventing COVID-19 Spread in Healthy Subjects:

Summary: This study will evaluate in a PH I/II trial in healthy volunteers the safety and tolerability of PVP-I nasal swabs daily application. The intent is to follow with a PH III randomized controlled clinical trial to assess the capacity for PVP-I nasal swabs to mitigate the transmission of respiratory viruses specifically COVID 19.

DETAILED DESCRIPTION:
Specific Aim 1: Evaluate toxicity and tolerability of PVP-I nasal swabs Specific Aim 2: Investigate the dosing of PVP-I nasal swabs.

Hypothesis 1: PVP-I nasal swabs have a low toxicity, low side effect profile, and high tolerability with daily use.

Hypothesis 2: Twice a day dosing for six weeks will prove safe in this subject population.

Healthy volunteers living in the Boston area between the ages of 18 and 70 years old will be recruited for participation in this study.

Consenting subjects will undergo baseline testing to confirm participants eligibility for this trial. As mentioned above, the target for enrollment is 50 subjects, so it is anticipated that approximately 75 subjects will be recruited, consented, and screened/tested, with about 25 of those subjects being either ineligible after testing or unable to complete the full 12 weeks of the trial. Subjects will apply 3M's PVP-I nasal swabs either once (control group) or twice (treatment group) per day, depending on the group that participants are randomized into. Subjects will apply the nasal swabs daily for six weeks with weekly symptom assessments and testing. After subjects cease nasal swab application, participants will return after another six weeks (i.e. 12 weeks after participants first nasal swab application) for a final round of testing and symptom assessment. Subjects will not need to pay for any nasal swabs or visits during this trial - all study-related items and visits will be covered by the sponsor. Subjects will also be remunerated with up to 100 dollars in gift certificates if participants complete the study and attend the check-ins (50 dollar certificate for completing baseline visit and 50 dollar certificate for coming in at 12 weeks).

Baseline screening will assess the overall health of the subject, confirm that participants have no underlying cardiac or thyroid conditions, participants are not pregnant (serum hCG testing will confirm this) nor intend to conceive during the course of this trial, and that participants are not experiencing any symptoms of COVID-19 (e.g. coughing, fever, shortness of breath). Further, testing will include thyroid stimulating hormone (TSH), thyroid peroxidase (TPO) antibody, serum human chorionic gonadotropin (hCG; to test for pregnancy), urine iodine, and COVID-19 mRNA (for the presence of an active virus) and antibody (as evidence for previous COVID-19 infection). Some of these tests will be administered weekly, at baseline only, at six weeks, or at 12 weeks. All research-related phlebotomy for this study will take place at BWH clinical research phlebotomy labs, such as the Clinical Trials Hub at 60 Fenwood Road or the Clinical Trials Center at 15 Francis Street. Again, all tests are covered by study funding and subjects will never be charged for them.

Once subjects' test results are returned and participants are deemed eligible for the study, participants will meet with the investigator in a clinical exam room (with masks and 6 feet social distance), and the investigator will demonstrate how to apply the nasal swabs so that the subject can continue to apply the swabs by themselves for the duration of the study. The investigator will assure that the subject has learned how to apply the nasal swab correctly and safely and that the subject understands the importance of daily, regimented application. Alternatively, if the subject would prefer to minimize in-person contact with others, participants can obtain the study drug from the investigator or study staff and learn how to apply the swabs through a Zoom meeting. Further, a video detailing these instructions will be sent to subjects with detailed application instructions.

Subjects will also be given a questionnaire to fill out at each weekly check-in, which will assess any side effects participants may be experiencing related to this drug (questionnaire is attached to this IRB submission on Insight). Questions will be focused on symptoms of hyperthyroidism (e.g. palpitations, tremulousness, weight loss, irritability) and hypothyroidism (e.g. fatigue, weight gain, sluggishness, hair loss). Subjects will also be informed at the time of enrollment that if participants start experiencing any troubling side effects, participants should stop applying swabs and alert study staff or an investigator of these side effects as soon as participants can. If this happens, or if a subject's test results reveal markers that are outside of reference ranges, participants will be withdrawn from the study and investigators will explain why participants are being withdrawn. Investigators will closely monitor the safety of patients and alert the FDA and the BWH IRB if any adverse events occur. However, given the proven safety of PVP-I and the weekly testing and assessments the investigators are conducting, the investigators do not anticipate that any adverse events will occur.

The overall study, from initiation and patient recruitment to data analysis and synthesis of a detailed report is anticipated to take six months.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy volunteers from the Boston community
2. 18-70 years of age
3. In good health, without thyroid or cardiac disease, without symptoms of COVID-19*
4. Normal baseline TSH

Exclusion Criteria:

1. History of thyroid or cardiac disease
2. Current BWH employee
3. Allergy or hypersensitivity to iodine
4. Positive COVID-19 mRNA or antibody test
5. Participation in any other investigational study or drug trial in which receipt of an investigational study drug occurred within 30 days prior to enrollment in this study
6. Women who are pregnant or attempting to conceive
7. Men who are attempting to conceive with their partner

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-08 (Estimated); Primary Completion 2021-02 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by self reporting, metabolic and endocrine metrics | follow up until 12 weeks
  Safety and tolerability assessment of PVP-I nasal swabs with 5% PVP-I with 0.5% available iodine will be ascertained using weekly measurements of iodine metabolism, thyroid function testing and self reporting of symptoms.

SECONDARY OUTCOMES:
Number of participants with dose dependent side effects determined by self reporting diaries, thyroid and metabolic testing | follow up until 12 weeks
  Investigate the dosing of PVP-I nasal swabs twice a day for six weeks with follow up to 12 weeks. The investigators will assess for iodine dose dependent side effects, changes in thyroid functions or iodine clearance.

IPD SHARING:
Plan to Share IPD: No
Anonymized, de-identified aggregate data that cannot be traced or linked to the participant.